CLINICAL TRIAL: NCT06513988
Title: Application of MI-BCI Combined With tDCS in Early Rehabilitation After Anterior Cruciate Ligament Reconstruction Monitored by Resting-stage fMRI: the First Case Report
Brief Title: Application of MI-BCI Combined With tDCS in Early Rehabilitation After Anterior Cruciate Ligament Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Chongwen Zuo, Principal Investigator, Air Force Military Medical University, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Air Force Medical Center
Record Dates: First submitted 2024-07-16; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Anterior Cruciate Ligament Injuries
Keywords: fMRI; MI-BCI; tDCS; after anterior cruciate ligament
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MI-BCI combined with tDCS (Experimental): The MI-BCI combined with tDCS treatment was performed five days per week (in the late afternoon)
  Interventions: Device: MI-BCI combined with tDCS treatment

INTERVENTIONS:
Device: MI-BCI combined with tDCS treatment — The treatment intervention was carried out in an independent and quite room and included following steps: During the MI-BCI based training, MI of leg flexion and extension training was first performed 10 times to accurate the training threshold, and then later in the formal BCI training, if the attention was reached the threshold, functional electrical stimulator was trigger to stimulate the corresponding muscle to execute the actual action. Additionally, the patient was given a brief training about how to operate tDCS device until he felt comfortable using it, and then asked to show and give feedback to the researcher. For motor function and pain improvement, tDCS is typically delivered with the anode electrode placed over the primary motor cortex (M1), and the cathode over the supraorbital area (SO) to trigger neuroplastic changes[5]. The MI-BCI combined with tDCS treatment was performed five days per week (in the late afternoon), and MI-BCI training for 30min.

SUMMARY:
To recover lower-limb motor function is a primary goal for rehabilitation after anterior cruciate ligament (ACL) reconstruction. Although quantitative testing and questionnaire evaluation provide a lot of valuable information, while functional magnetic resonance imaging (fMRI) provides a powerful method to assess functional connectivity (FC) involved in motor function recovery before and after receiving a novel combined rehabilitation training. However, our understanding of the FC changes during early rehabilitation after ACL reconstruction is partial and incomplete.

DETAILED DESCRIPTION:
ACL has become one of the most common and easily damaged knee ligaments in sports and military training affecting young and active people. The extensive interest in ACL ruptures is related to the subsequent articular degeneration and severe dysfunction, resulting in skeletal muscle functional limitations not only in athletics but also in daily living. Thus, restoring lower limb motor function and stability has become the primary goal after ACL reconstruction (ACLR). Moreover, the newest study has indicated that increased neural activity may reflect central neuroplastic strategies to preserve motor functionality after ACLR[1]. Postsurgical rehabilitation guidelines for the orthopedic clinician recommended a common treatments for ACLR patients[2]; however, because of long time consuming and poor compliance, which are difficult to get patient recognition, it is very urgent to find a safe, effective and easy conduct and alternative therapy. Transcranial direct-current stimulation (tDCS) is a non-invasive technique of brain stimulation that has potential for clinical utility in neurorehabilitation, and could improve the lower excitability, muscle strength and dynamic balance by acting on the primary motor cortex[3]. For another, motor imagery based brain-computer interface (MI-BCI) based neuro rehabilitation paradigms have emerged as a novel iatrotechnics on motor function and brain function recovery[4]. However, it is little explored whether the clinical application of MI-BCI therapy combined with tDCS could be effective for early rehabilitation after ACLR patients. This case report would explore the efficacy and neuromechanism for the ACLR patient treated with MI-BCI training combined with tDCS. BOLD-fMRI was performed before and after four weeks' treatment.

ELIGIBILITY:
Inclusion Criteria:

* Duration of anterior cruciate ligament injury: 3-12 months
* Must bet acceptted anterior cruciate ligament reconstruction

Exclusion Criteria:

* The affected limb has severe ligament and meniscus damage
* Contralateral lower extremity sports injury
* Other medical conditions, such as severe disc herniation, are not eligible for the test

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2024-05-06 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
resting-stage fMRI | before and after 4 weeks
  Resting-stage fMRI images data acquisition was carried out in the Air Force Medical Center with a 3.0T MRI scanner (GE Discovery MR750, USA) using the echo planar imaging (BOLD) sequence for 6 min each time (TR/TE = 2000 ms/30 ms, matrix 64 × 64, FOV = 220×220mm2, number of slices = 36) with contiguous 3 mm slice thickness providing whole brain coverage. In addition, a series of anatomical images were also obtained during the first imaging session using T1-weighted 3D TFE sequence with 1×1×1mm resolution
IKDC | before and after 4 weeks
  The IKDC score is a subjective knee assessment scale used to assess the level of knee function and severity of symptoms. The functional status of the knee joint is assessed by summing the scores for each item, converting the scores to a scale of 0 to 100

CONTACTS AND LOCATIONS:
Overall Officials: Chongwen Zuo, Doctoral, Principal Investigator — Air Force Medical Center of Chinese PLA
Locations (1):
- Air Force Medical Center of PLA, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR